CLINICAL TRIAL: NCT02370680
Title: Durability of Antiplatelet Effect of a Novel Extended-Release Formulation of Acetylsalicylic Acid, Durlaza in CVD (Cardiovascular Disease) Patients at Risk of High Platelet Turnover
Brief Title: Length of Effect of Extended Release Aspirin on Platelets in Patients With Diabetes and Heart Disease
Acronym: DURATION
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: New Haven Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NHP-ASP-102
Record Dates: First submitted 2015-02-11; First posted 2015-02-25 (Estimated); Last update posted 2015-08-06 (Estimated); Status verified 2015-08

CONDITIONS: Cardiovascular Disease
Keywords: Antiplatelet; Antiplatelet therapy; platelet turnover; high platelet turnover; platelet aggregation; cardiovascular disease; coronary artery disease; diabetes mellitus
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Artery Disease; Diabetes Mellitus | interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Durlaza™, 1 capsule (Experimental): Aspirin run-in, followed with Durlaza™, one capsule QD (quaque die), for 14 ± 4 days and an in-patient visit
  Interventions: Drug: Aspirin; Drug: Durlaza™
- Durlaza™, 2 capsules (Experimental): in a rollover with 10 subjects from the first arm, an aspirin run-in, followed by Durlaza™, two capsules QD, for 14 ± 4 days and an in-patient visit
  Interventions: Drug: Aspirin; Drug: Durlaza™

INTERVENTIONS:
Drug: Aspirin — steady-state run-in prior to Durlaza treatment
  Other Names: Bayer aspirin
Drug: Durlaza™ — comparison of different numbers of capsules

SUMMARY:
This study is being conducted to evaluate the safety and the length of effect on platelet build-up in the arteries of Durlaza™ as compared to immediate-release Bayer® aspirin 81 mg or subject's current aspirin 81 mg of choice in patients who have Type 2 diabetes mellitus and cardiovascular disease or multiple risk factors of developing cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-lactating, non-pregnant female subjects
* A history of Type 2 Diabetes and with history of at least one of the following: Coronary Artery Disease, Peripheral Vascular Disease, or Ischemic Stroke, along with at least 2 CVD risk factors (obese, smoker, ≥ 55 years of age, prior thrombotic event)

Exclusion Criteria:

* Sensitivity to aspirin or any NSAID (nonsteroidal antiinflammatory drug),
* Evidence of uncontrolled or unstable cardio- or cerebrovascular disorder,
* Presence of uncontrolled or chronic medical illness, GI disorder or surgery leading to impaired drug absorption, clinically significant abnormal baseline ECG, history of hepatitis, malignancy within the past five years, or HIV, history of alcohol or drug abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2015-02; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
change in platelet aggregation | During the 26-hour hospital stays, outcomes will be measured at various timepoints

SECONDARY OUTCOMES:
Reactive Hyperemia Index | During the 26-hour hospital stays, outcomes will be measured at various timepoints
Safety as measured by the number and system class of adverse events reported in each treatment arm | participants are followed for approximately 40 to 65 days once they start study medication

OTHER OUTCOMES:
Serum Thromboxane | During the 26-hour hospital stays, outcomes will be measured at various timepoints
urinary metabolites of prostacyclin and thromboxane | During the 26-hour hospital stays, outcomes will be measured at various timepoints

CONTACTS AND LOCATIONS:
Overall Officials: Paul Gurbel, MD, Principal Investigator — Platelet Thrombosis Research, LLC
Locations (1):
- Platelet and Thrombosis Research, LLC, Baltimore, Maryland, United States